CLINICAL TRIAL: NCT05762952
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate Microvascular Disease After 12 Weeks of Therapy With Sodium-glucose Co-transporter 2 Inhibitor Compared to Placebo in Symptomatic Women With Non-obstructive Coronary Artery Disease
Brief Title: Effect of Dapagliflozin on Microvascular Function in Women With Symptoms of Coronary Artery Disease
Acronym: SMILE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Patricia Rodriguez Lozano, Assistant Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR220123
Record Dates: First submitted 2023-01-09; First posted 2023-03-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — dapagliflozin; Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy will manage the randomization of study participants. Assignments will not be unmasked until all outcomes have been assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10mg oral tablet.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo (Placebo Comparator): Placebo matching tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Once daily oral dapagliflozin 10mg
  Other Names: active drug
  Arms: Dapagliflozin
Drug: Placebo — Placebo capsules formulated by pharmacy to be indistinguishable from active drug
  Other Names: Placebo matching tablet
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test the effects of a drug (in the drug class called sodium-glucose cotransporter 2 inhibitors) in women who have symptoms of ischemic heart disease. The main questions the study aims to answer are:

Does blood flow in the heart improve with study drug?

Participants will be randomly assigned to a 12-week course of the study drug, dapagliflozin 10mg, or placebo. Blood flow in the heart will be assessed using stress cardiac magnetic resonance imaging at baseline and 12 weeks. The researchers will compare the results from the two groups.

DETAILED DESCRIPTION:
This single-center clinical investigation is a randomized, double-blind, placebo controlled trial of dapagliflozin in women who have symptoms of myocardial ischemia but in whom obstructive coronary artery disease has been ruled out by testing within 2 years.

Aim: Determine whether dapagliflozin improves coronary blood flow in women.

Participants will be randomly assigned to a 12-week course of dapagliflozin 10mg oral or placebo. Participants will complete study assessments at baseline, 6 weeks of treatment, and 12 weeks of treatment. Peak myocardial blood flows at rest and with pharmacological stress will be assessed using cardiac magnetic resonance imaging at baseline and 12 weeks. Symptom surveys and lab work will be collected at baseline, 6 weeks, and 12 weeks of treatment. Participants will be closely monitored throughout study participation for adverse events. Results will be captured in a database and published in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent.
* Signs and symptoms of suspected ischemia that prompted referral for further evaluation by cardiac catheterization or coronary computed tomography within two years of consent.
* No evidence of obstructive epicardial coronary artery disease (stenosis >50%) of a major epicardial vessel (>3mm) or a fractional flow reserve >0.80 by invasive catheterization or coronary computed tomography. (Participants who have not undergone cardiac catheterization or coronary angiogram within the last 2 years for their clinical care will be screened with computed angiogram of the coronary arteries to confirm eligibility).
* Estimated glomerular filtration rate ≥30ml/min/1.73m2 at enrollment
* For subjects having a history of type 2 diabetes mellitus: approval of diabetes care/prescribing provider

Exclusion Criteria:

* History of non-ischemic cardiomyopathy with left ventricular ejection fraction <40% or hypertrophic cardiomyopathy.
* History of congestive heart failure, severe pulmonary disease, liver disease
* History of Acute coronary syndrome within previous 30 days
* Stroke within the last 180 days or intracranial hemorrhage at any time.
* Severe Valvular disease
* Life expectancy <3 years, due to non-cardiovascular comorbidity.
* Pregnancy or women who are breast-feeding
* Type 1 diabetes mellitus
* History of diabetic ketoacidosis in subjects with Type 2 Diabetes Mellitus
* Symptomatic hypotension or systolic blood pressure <95 mmHg on 2 consecutive measurements
* Active malignancy requiring treatment at the time of visit
* Severe, unstable, or rapidly progressing renal disease at the time of randomization
* History of recurrent urinary tract, bladder, or kidney infections

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial perfusion reserve | Baseline and after 12 weeks of treatment
  Myocardial microvascular perfusion, defined as myocardial perfusion reserve as assessed by stress cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Rodriguez-Lozano, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No